CLINICAL TRIAL: NCT00079365
Title: A Randomized Trial Comparing 5-Fluorouracil, External Beam Radiation, and Gemcitabine With or Without P Radiopharmaceutical Therapy As A First Line Therapy in Patients With Locally/Regionally Advanced Non-Resectable Adenocarcinoma of the Pancreas
Brief Title: Fluorouracil, External-Beam Radiation Therapy, and Gemcitabine With or Without Brachytherapy Using Phosphorus P32 in Treating Patients With Locally or Regionally Advanced Unresectable Adenocarcinoma of the Pancreas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of South Florida (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000355400; USFPG-6034
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2005-05

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Brachytherapy; Phosphorus-32; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Radiation: brachytherapy
Radiation: phosphorus P32
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Fluorouracil may make the tumor cells more sensitive to radiation therapy. Brachytherapy uses radioactive material, such as phosphorus P32, placed directly into or near a tumor to kill tumor cells. Combining chemotherapy and external-beam radiation therapy with brachytherapy may kill more tumor cells.

PURPOSE: This randomized clinical trial is studying fluorouracil, gemcitabine, external-beam radiation therapy, and brachytherapy using phosphorus P32 to see how well they work compared to fluorouracil, gemcitabine, and external-beam radiation therapy in treating patients with locally or regionally advanced unresectable adenocarcinoma of the pancreas (pancreatic cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients with locally or regionally advanced unresectable adenocarcinoma of the pancreas treated with fluorouracil, external beam radiotherapy, and gemcitabine with vs without brachytherapy with phosphorus P32 suspension.

Secondary

* Compare time to disease progression, tumor response rate, and physical performance in patients treated with these regimens.
* Compare the safety and tolerability of these regimens in this patient population.
* Compare duration of response and time to treatment failure in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive phosphorus P32 suspension percutaneously under CT guidance on day 0 and at months 1, 2, 6, 7, and 8. Patients receive fluorouracil IV continuously on days 1-5 of weeks 1-6. Patients concurrently undergo external beam radiotherapy 5 days a week on weeks 1-6. At the completion of radiotherapy, patients receive gemcitabine IV over 30 minutes once weekly for 7 weeks. After a 1-week rest, patients then receive gemcitabine IV over 30 minutes once weekly for 3 weeks. Treatment repeats every 28 days.
* Arm II: Patients receive fluorouracil and gemcitabine and undergo external beam radiotherapy as in arm I.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 80 patients (40 per treatment arm) will be accrued for this study within 24-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Locally or regionally advanced disease
* Unresectable disease defined by the following:

  * Invasion into a major vascular structure determined preoperatively by a CT scan, angiogram, or CT portogram or intraoperatively by surgeon
  * Severe comorbidities precluding operation, such as congestive heart failure, coronary artery disease, or chronic obstructive pulmonary disease
* Bidimensionally measurable disease by CT scan
* No recurrent disease
* No previously resected pancreatic cancer
* No tumors of the pancreas not ductal in origin (e.g., islet cell tumors, lymphoma, or sarcoma)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count: ≥ 1,500/mm^3
* Platelet count ≥ 50,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 5 times ULN
* Alkaline phosphatase < 5 times ULN
* Albumin ≥ 2.5 mg/dL

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* See Disease Characteristics

Pulmonary

* See Disease Characteristics

Other

* No other malignancy within the past 5 years except curatively resected basal cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or early stage prostate cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for pancreatic adenocarcinoma

Surgery

* See Disease Characteristics

Other

* No prior chromic phosphate P32 suspension (Phosphocol®)
* At least 4 weeks since prior cytotoxic therapy for pancreatic adenocarcinoma
* At least 4 weeks since prior investigational anti-tumoral agents
* No other concurrent investigational agents
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rosemurgy, MD, Study Chair — University of South Florida
Locations (1):
- USF Physician's Group, Tampa, Florida, United States